CLINICAL TRIAL: NCT05436847
Title: Effects of Proprioceptive Training in Addition to Routine Physical Therapy on Gross Motor Function in Children With Spastic Quadriplegic Cerebral Palsy: A Randomized Control Trial
Brief Title: Effects of Proprioceptive Training With Routine PT on Gross Motor Function in Spastic Quadriplegic CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/831-VI/2021
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy
Keywords: : Spastic Quadriplegia, Cerebral palsy; Proprioceptive training, Somatosensory input
MeSH Terms: conditions — Cerebral Palsy; Quadriplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): NDT- age appropriate Transitions (age appropriate) Milestones training (age appropriate) Proprioceptive Input- age appropriate (Pushups Static quadruped, squat sitting, trampoline, hopping etc. With weights and splints for joint to joint approximation)
  Interventions: Other: Proprioceptive Training
- Group B (Active Comparator): NDT- age appropriate Transitions (age appropriate) Milestones training (age appropriate)
  Interventions: Other: Routine Physical Therapy

INTERVENTIONS:
Other: Proprioceptive Training — Proprioceptive Training using increased joint to joint approximation through ankle weights and joint splints.
  Arms: Group A
Other: Routine Physical Therapy — Neurodevelopmental treatment- age appropriate
  Arms: Group B

SUMMARY:
The proprioceptive training with a therapy regime enhances the body's somatosensory input that in result changes the body to be more functional in different types of interactions. This study is dedicated to finding out how much proprioception training is helpful in gross motor function level improvement and enhances functional activities of CP children

DETAILED DESCRIPTION:
Proprioception plays an important role in the correct execution of efferent motor performance as 70% of cerebral palsy population have deficit in receiving somatosensory signals3. Tradition physical therapy exercises including strengthening followed by stretching etc. should be reviewed and the therapy must be more oriented to overall individual growth and development31. There is a need to push the cerebral palsy population to be exercised with proprioceptive stimulation for their maximum participation in the activities of daily life including both personal and social aspects. The proprioceptive training with a therapy regime enhances the body's somatosensory input that in result changes the body to be more functional in different types of interactions. This study is dedicated to finding out how much proprioception training is helpful in gross motor function level improvement and enhances functional activities of CP children.

ELIGIBILITY:
Inclusion Criteria:

* Children with the diagnosis of Cerebral Palsy (Spastic quadriplegia)
* Ages of 1 to 5 years
* Both males and females
* Alert and responsive to verbal and non-verbal commands
* Modified Ashworth Sale grade 1 to 2
* Gross Motor Function Classification System level 1V and V

Exclusion Criteria:

* Children under the botox treatment for tone management (botulinum injections)
* Diagnosed with any disease other than spastic quadriplegic cerebral palsy i.e. congenital heart defects, epilepsy, recurrent pneumonia, skin infections etc.
* Children underwent any surgery i.e. tenotomy (tendon release), recent heart surgery,
* Recent fracture and subluxation/dislocation due to fall or poor handling
* Any contracture or deformity on upper extremities, lower extremities and spine i.e. flexion contractures, club foot, scoliosis

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function | 9 months
  Gross Motor Function Classification System (GMFCS) is a 5-level clinical classification system that describes the gross motor function of people with cerebral palsy on the basis of self-initiated movement abilities. Higher scores indicate better improvement in gross motor functions.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Jawad, MSPTN, Principal Investigator — University of Lahore
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No